CLINICAL TRIAL: NCT05866575
Title: Prediction of the Therapeutic Response in Depression Based on an Early Neuro-computational Modeling Assessment of Motivation
Brief Title: Prediction of the Therapeutic Response in Depression Based on Neuro-computational Modeling Assessment of Motivation
Acronym: STRATIDEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D20-P059
Record Dates: First submitted 2022-11-15; First posted 2023-05-19 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Vortioxetine

STUDY DESIGN:
Intervention Model Description: Randomization and introduction of the new antidepressant will occur immediately after V1. Patients will receive an antidepressant as monotherapy after randomization between two strategies: escitalopram and vortioxetine. To maximize acceptability by referring psychiatrists, dosage and co-prescriptions will be at the discretion of the psychiatrist in charge, but the allocated treatment will not be changed for 4 weeks (until V3).
  After 4 weeks, the treatment can be adapted by the refeering psychiatrist exactly as if the patient had not been included in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- escitalopram strategy (Other): The strategy will not be modified for a period of 4 weeks. Dosage adjustment and co-prescriptions will be at the discretion of the refeering psychiatrist.
  Interventions: Other: escitalopram
- vortioxetine strategy (Other): The strategy will not be modified for a period of 4 weeks. Dosage adjustment and co-prescriptions will be at the discretion of the refeering psychiatrist.
  Interventions: Other: vortioxetine

INTERVENTIONS:
Other: escitalopram — Patients will receive an antidepressant strategy : escitalopram. The strategy will not be modified for a period of 4 weeks. Dosage adjustment and co-prescriptions will be at the discretion of the refeering psychiatrist. After 4 weeks, the strategy can be adapted by the refeering psychiatrist exactly as if the patient had not been included in the trial.
  Arms: escitalopram strategy
Other: vortioxetine — Patients will receive an antidepressant strategy : vortioxetine. The strategy will not be modified for a period of 4 weeks. Dosage adjustment and co-prescriptions will be at the discretion of the refeering psychiatrist. After 4 weeks, the treatment strategy can be adapted by the refeering psychiatrist exactly as if the patient had not been included in the trial.
  Arms: vortioxetine strategy

SUMMARY:
This study aims to better understand the mechanisms of action of antidepressants, but also the neural correlates of motivation deficits. One hundred patients with a moderate to severe major depressive episode will be enrolled in this prospective multicenter study. The objective will be to predict the therapeutic response to two first-line antidepressants on the basis of an early neurocomputational assessment of motivation. Antidepressant treatment will be administered as monotherapy after randomization between two drugs: escitalopram and vortioxetine. Patients will undergo six visits and follow-up for one year. The investigators will combine computer modeling and functional MRI to identify motivational deficits and elucidate their brain correlates before initiation, after 7 days and after 6 months of treatment. 36 healthy volunteers will also be included to allow comparison with patients with depression. They will not receive any treatment.

DETAILED DESCRIPTION:
One hundred patients with a moderate to severe major depressive episode will be enrolled in this prospective multicenter study. Six visits will be scheduled within a year:

* V0 (inclusion visit): verification of inclusion and exclusion criteria, information, and consent.
* V1 (before randomization - baseline state):

  * Clinical evaluation using validated questionnaires for the severity of depression, quality of life, anhedonia, apathy, and cognitive dysfunction.
  * Neuro-cognitive evaluation using a battery of tests to explore motivation, emotion processing, belief construction, and their updating. Part of the tests will be performed during the functional MRI session.
  * Structural (anatomical) and functional MRI, ASL.
  * Blood samples.
  * Randomization and introduction of the new antidepressant will occur immediately after V1. To maximize acceptability by referring psychiatrists, dosage and co-prescriptions will be at the discretion of the psychiatrist in charge, but the assigned treatment will not be changed for 4 weeks (until V3).
* V2 (7 days after the beginning of the new antidepressant - 'early response visit'):

  o Similar to V1.
* V3 (28 days after the beginning of the new antidepressant - 'conventional response visit'):

  * Clinical evaluation using validated questionnaires for the severity of depression, quality of life, anhedonia, apathy, and cognitive dysfunction.
  * Blood samples
* V4 (6 months after the beginning of the new antidepressant - 'remission visit'):

  * Clinical evaluation using validated questionnaires for the severity of depression, quality of life, anhedonia, apathy, and cognitive dysfunction.
  * Cognitive evaluation using a battery of tests to explore motivation, emotion processing, belief construction, and their updating.
  * Structural (anatomical) MRI, ASL
  * Blood samples
* V5 (one year after the beginning of the new antidepressant - 'functional remission visit'):

  * Clinical evaluation using validated questionnaires for the severity of depression, quality of life, anhedonia, apathy, and cognitive dysfunction.

    36 healthy volunteers without a history of neurologic or psychiatric disorder, matched for age, gender, and education will be included. They will perform V0-V2 (without MRI and blood sample at V2). Healthy volunteers will not receive any treatment as part of the research.

ELIGIBILITY:
Patients with major depressive disorder

Inclusion Criteria:

* Meeting DSM-5 criteria for major depressive disorder (single or recurrent episodes)
* With a MADRS score >= 24
* For which a new line of treatment is needed
* No previous line of antidepressant for this episode or wash-out long-enough to avoid carry-over effects
* Valid health care insurance

Exclusion Criteria:

* Treatment-resistant depression (defined as insufficient response despite at least 2 trials of antidepressant prescribed at adequate dose and duration)
* Subjects with a trial of escitalopram and/or vortioxetine for the current episode, or with contra-indication to one of these two drugs
* Subjects with a diagnostic of persistent depressive disorder, bipolar disorder or schizophrenia, neurodeveloppemental disorder, unremitted substance abuse disorder other than tobacco, personality disorder severe enough to compromise the follow-up (based on investigator's appreciation).
* Subject with a history of neurological disorder: parkinson's disease, dementia
* Contraindications to MRI scanning: pregnancy, claustrophobia, metallic implants
* Pregnant or breastfeeding women
* involuntary hospitalisation and legal protection measures

Healthy volunteers

Inclusion Criteria:

- Valid health care insurance

Exclusion Criteria:

* Subjects with a diagnostic of persistent depressive disorder, bipolar disorder or schizophrenia, neurodeveloppemental disorder, unremitted substance abuse disorder other than tobacco, personality disorder severe enough to compromise the follow-up (based on investigator's appreciation).
* Subject with a history of neurological disorder: parkinson's disease, dementia
* Contraindications to MRI scanning: pregnancy, claustrophobia, metallic implants
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of the therapeutic response (MADRS score) 28 days after the introduction of the antidepressant strategy (V3) based on the early changes (differences between V1 and V2) of the computational phenotype of depressed patients. | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant) and V3 (after 28 days of antidepressant)
  The therapeutic response will be measured with the Montgomery-Asberg Depression Rating Scale (MADRS). The MADRS is a 10- item scale widely used in depression research to assess the severity of depression. Response will be defined by a score divided by 2 compared to baseline MADRS score, while remission will be defined by a score < 7 (symptom absent) 28 days after the initiation of the antidepressant strategy.
  The "computational phenotype" is the outcome of the computationnal analysis of behavior. It is expressed in abstract unit. The change in computationnal phenotype between V1 and V2 will be entered in logistic regression aiming to predict clinical response at 28 days, measured with the MADRS score.

SECONDARY OUTCOMES:
Prediction of the therapeutic response (MADRS score) 28 days after the introduction of the antidepressant strategy (V3) based on the early changes (differences between V1 and V2) of the neuro-computational phenotype of depressed patients | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant) and V3 (after 28 days of antidepressant)
  Same than outcome 1 but using brain imaging on top of behavior (neurocomputational modeling) to predict clinical response.
Prediction of the therapeutic response (MADRS score) 28 days after the introduction of the antidepressant strategy (V3) based on the initial (baseline state- V1) neuro-computational phenotype of depressed patients | Baseline state (before the start of antidepressant strategy), and V3 (after 28 days of antidepressant)
  Same than Outcome 2 but using only V1 instead of the change between V1 and V2 to predict clinical response.
Prediction of long-term remission (V4) based on the early changes (differences between V1 and V2) of the neuro-computationnal phenotype of depressed patients | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant), V4 (6 months after the start of antidepressant)
  Same than Outcome 2 but to predict clinical remission at V4 instead of clinical response at V3.
Prediction functional remission (V5) based on the early changes (differences between V1 and V2) of the neuro-computationnal phenotype of depressed patients | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant), V5 (1 year after the start of antidepressant)
  Same than Outcome 2 but to predict functional remission at V5 instead of clinical response at V3.
Prediction of relapse at one year (V5) based on the computationnal phenotype of remitted patients at 6 months (V4). | V4 (6 months after the start of antidepressant), V5 (1 year after the start of antidepressant)
  Same than Outcome 1 but using computational phenotype at V4 to predict predict functional remission at V5.
Description of the motivational deficit of depressed patients at baseline (V1). | Baseline state (before the start of antidepressant strategy)
  Comparison of the computational phenotype of patients with depression and healthy volunteers at V1.
Description of the neural correlates of motivation deficits of depressed patients at baseline (V1). | Baseline state (before the start of antidepressant strategy)
  Comparison of the brain functional statistical maps of patient with depression and healthy volunteers at V1.
Description of the evolution of motivation deficit of depressed patients after one week of antidepressant treatment | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant)
  Comparison of the computational phenotype of patients with depression at V1 and V2.
Description of the evolution of the neural correlates of motivation deficits after one week of antidepressant treatment | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant)
  Comparison of the brain functional statistical maps of patient with depression at V1 and V2.
Description of the evolution of motivation deficit of depressed patients at 6 months | Baseline state (before the start of antidepressant strategy), V4 (6 months after the start of antidepressant)
  Comparison of the computational phenotype of patients with depression at V1 and V4.
Description of the evolution of the structural neural correlates of depression after 6 months of treatment | Baseline state (before the start of antidepressant strategy), V4 (6 months after the start of antidepressant)
  Comparison of the structural brain imaging of patients with depression at V1 and V4.
Description of the evolution of the functional neural correlates of depression after 6 months of treatment | Baseline state (before the start of antidepressant strategy) V4 (6 months after the start of antidepressant)
  Comparison of the function brain imaging (ASL) of patients with depression at V1 and V4.
Construction of a bio-bank | Baseline state (before the start of antidepressant strategy), V2 (after 7 days of antidepressant) and V3 (after 28 days of antidepressant), V4 (6 months after the start of antidepressant)
  Serum tubes will be drowned along the study (V1, V2, V3 and V4 for patients - V1 for healthy volunteers) prepared and stored.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Groupe hospitalo-universitaire de Grenoble Alpes, La Tronche, Isère
  - Centre hospitalier Universitaire de Lille, Lille, Nord
  - Centre hospitalier Universitaire de Saint-Etienne, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Groupe hospitalo-universitaire Assistance Publique, hôpital Pitié Salpêtrière - Hôpitaux de Paris Sorbonne Université, Paris
  - - Groupe hospitalo-universitaire Paris Psychiatrie et Neurosciences, Paris

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from medical visits (clinical informations, biological assessments, cognitive data) and brain MRIs will be kept, coded and archived for a period of two years after the last publication of the research results or until the final research report is signed. These can be used later for collaborative research (academic and/or industrial partners) in the European Union (EU) and/or abroad exclusively for scientific purposes.
  In case of transfer of the anonymized database resulting from this research abroad (outside the EU), the sponsor undertakes to ensure a level of security equivalent to French or European Union law.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data obtained from medical visits (clinical informations, biological assessments, neurocognitive data)and brain MRIs will be kept, coded and archived for a period of two years after the last publication of the research results or until the final research report is signed.
Access Criteria: The data can be used for collaborative research (academic and/or industrial partners) in the European Union (EU) and/or abroad exclusively for scientific purposes.
  In case of transfer of the anonymized database resulting from this research abroad (outside the EU), the sponsor undertakes to ensure a level of security equivalent to French or European Union law.

REFERENCES:
- [Background] Bauer M, Pfennig A, Severus E, Whybrow PC, Angst J, Moller HJ; World Federation of Societies of Biological Psychiatry. Task Force on Unipolar Depressive Disorders. World Federation of Societies of Biological Psychiatry (WFSBP) guidelines for biological treatment of unipolar depressive disorders, part 1: update 2013 on the acute and continuation treatment of unipolar depressive disorders. World J Biol Psychiatry. 2013 Jul;14(5):334-85. doi: 10.3109/15622975.2013.804195. Epub 2013 Jul 3. PMID 23879318
- [Background] Lam RW, Kennedy SH, Grigoriadis S, McIntyre RS, Milev R, Ramasubbu R, Parikh SV, Patten SB, Ravindran AV; Canadian Network for Mood and Anxiety Treatments (CANMAT). Canadian Network for Mood and Anxiety Treatments (CANMAT) clinical guidelines for the management of major depressive disorder in adults. III. Pharmacotherapy. J Affect Disord. 2009 Oct;117 Suppl 1:S26-43. doi: 10.1016/j.jad.2009.06.041. Epub 2009 Aug 11. PMID 19674794
- [Background] Uher R, Perlis RH, Henigsberg N, Zobel A, Rietschel M, Mors O, Hauser J, Dernovsek MZ, Souery D, Bajs M, Maier W, Aitchison KJ, Farmer A, McGuffin P. Depression symptom dimensions as predictors of antidepressant treatment outcome: replicable evidence for interest-activity symptoms. Psychol Med. 2012 May;42(5):967-80. doi: 10.1017/S0033291711001905. Epub 2011 Sep 20. PMID 21929846
- [Background] Pessiglione M, Vinckier F, Bouret S, Daunizeau J, Le Bouc R. Why not try harder? Computational approach to motivation deficits in neuro-psychiatric diseases. Brain. 2018 Mar 1;141(3):629-650. doi: 10.1093/brain/awx278. PMID 29194534
- [Background] Clery-Melin ML, Schmidt L, Lafargue G, Baup N, Fossati P, Pessiglione M. Why don't you try harder? An investigation of effort production in major depression. PLoS One. 2011;6(8):e23178. doi: 10.1371/journal.pone.0023178. Epub 2011 Aug 10. PMID 21853083
- [Background] Mauras T, Masson M, Fossati P, Pessiglione M. Incentive Sensitivity as a Behavioral Marker of Clinical Remission From Major Depressive Episode. J Clin Psychiatry. 2016 Jun;77(6):e697-703. doi: 10.4088/JCP.15m09995. PMID 27337420
- [Background] Le Heron C, Plant O, Manohar S, Ang YS, Jackson M, Lennox G, Hu MT, Husain M. Distinct effects of apathy and dopamine on effort-based decision-making in Parkinson's disease. Brain. 2018 May 1;141(5):1455-1469. doi: 10.1093/brain/awy110. PMID 29672668
- [Background] Wardle MC, Treadway MT, Mayo LM, Zald DH, de Wit H. Amping up effort: effects of d-amphetamine on human effort-based decision-making. J Neurosci. 2011 Nov 16;31(46):16597-602. doi: 10.1523/JNEUROSCI.4387-11.2011. PMID 22090487
- [Background] Treadway MT, Buckholtz JW, Cowan RL, Woodward ND, Li R, Ansari MS, Baldwin RM, Schwartzman AN, Kessler RM, Zald DH. Dopaminergic mechanisms of individual differences in human effort-based decision-making. J Neurosci. 2012 May 2;32(18):6170-6. doi: 10.1523/JNEUROSCI.6459-11.2012. PMID 22553023
- [Background] Nutt D, Demyttenaere K, Janka Z, Aarre T, Bourin M, Canonico PL, Carrasco JL, Stahl S. The other face of depression, reduced positive affect: the role of catecholamines in causation and cure. J Psychopharmacol. 2007 Jul;21(5):461-71. doi: 10.1177/0269881106069938. Epub 2006 Oct 18. PMID 17050654
- [Background] Culpepper L. Escitalopram: A New SSRI for the Treatment of Depression in Primary Care. Prim Care Companion J Clin Psychiatry. 2002 Dec;4(6):209-214. doi: 10.4088/pcc.v04n0601. PMID 15014711
- [Background] Sanchez C, Asin KE, Artigas F. Vortioxetine, a novel antidepressant with multimodal activity: review of preclinical and clinical data. Pharmacol Ther. 2015 Jan;145:43-57. doi: 10.1016/j.pharmthera.2014.07.001. Epub 2014 Jul 9. PMID 25016186
- [Background] Fervaha G, Foussias G, Agid O, Remington G. Motivational and neurocognitive deficits are central to the prediction of longitudinal functional outcome in schizophrenia. Acta Psychiatr Scand. 2014 Oct;130(4):290-9. doi: 10.1111/acps.12289. Epub 2014 May 22. PMID 24850369
- [Background] Fervaha G, Foussias G, Takeuchi H, Agid O, Remington G. Motivational deficits in major depressive disorder: Cross-sectional and longitudinal relationships with functional impairment and subjective well-being. Compr Psychiatry. 2016 Apr;66:31-8. doi: 10.1016/j.comppsych.2015.12.004. Epub 2015 Dec 18. PMID 26995233
- [Background] Berwian IM, Wenzel JG, Collins AGE, Seifritz E, Stephan KE, Walter H, Huys QJM. Computational Mechanisms of Effort and Reward Decisions in Patients With Depression and Their Association With Relapse After Antidepressant Discontinuation. JAMA Psychiatry. 2020 May 1;77(5):513-522. doi: 10.1001/jamapsychiatry.2019.4971. PMID 32074255
- [Background] Schmidt L, Lebreton M, Clery-Melin ML, Daunizeau J, Pessiglione M. Neural mechanisms underlying motivation of mental versus physical effort. PLoS Biol. 2012 Feb;10(2):e1001266. doi: 10.1371/journal.pbio.1001266. Epub 2012 Feb 21. PMID 22363208
- [Background] Skvortsova V, Palminteri S, Pessiglione M. Learning to minimize efforts versus maximizing rewards: computational principles and neural correlates. J Neurosci. 2014 Nov 19;34(47):15621-30. doi: 10.1523/JNEUROSCI.1350-14.2014. PMID 25411490
- [Background] Pessiglione M, Schmidt L, Draganski B, Kalisch R, Lau H, Dolan RJ, Frith CD. How the brain translates money into force: a neuroimaging study of subliminal motivation. Science. 2007 May 11;316(5826):904-6. doi: 10.1126/science.1140459. Epub 2007 Apr 12. PMID 17431137
- [Background] Pessiglione M, Delgado MR. The good, the bad and the brain: Neural correlates of appetitive and aversive values underlying decision making. Curr Opin Behav Sci. 2015 Oct;5:78-84. doi: 10.1016/j.cobeha.2015.08.006. Epub 2015 Aug 24. PMID 31179377
- [Background] Palminteri S, Justo D, Jauffret C, Pavlicek B, Dauta A, Delmaire C, Czernecki V, Karachi C, Capelle L, Durr A, Pessiglione M. Critical roles for anterior insula and dorsal striatum in punishment-based avoidance learning. Neuron. 2012 Dec 6;76(5):998-1009. doi: 10.1016/j.neuron.2012.10.017. PMID 23217747
- [Background] Lebreton M, Jorge S, Michel V, Thirion B, Pessiglione M. An automatic valuation system in the human brain: evidence from functional neuroimaging. Neuron. 2009 Nov 12;64(3):431-9. doi: 10.1016/j.neuron.2009.09.040. PMID 19914190
- [Background] Vinckier F, Rigoux L, Oudiette D, Pessiglione M. Neuro-computational account of how mood fluctuations arise and affect decision making. Nat Commun. 2018 Apr 26;9(1):1708. doi: 10.1038/s41467-018-03774-z. PMID 29700303
- [Background] Stephan KE, Bach DR, Fletcher PC, Flint J, Frank MJ, Friston KJ, Heinz A, Huys QJM, Owen MJ, Binder EB, Dayan P, Johnstone EC, Meyer-Lindenberg A, Montague PR, Schnyder U, Wang XJ, Breakspear M. Charting the landscape of priority problems in psychiatry, part 1: classification and diagnosis. Lancet Psychiatry. 2016 Jan;3(1):77-83. doi: 10.1016/S2215-0366(15)00361-2. Epub 2015 Nov 11. PMID 26573970
- [Background] Stephan KE, Binder EB, Breakspear M, Dayan P, Johnstone EC, Meyer-Lindenberg A, Schnyder U, Wang XJ, Bach DR, Fletcher PC, Flint J, Frank MJ, Heinz A, Huys QJM, Montague PR, Owen MJ, Friston KJ. Charting the landscape of priority problems in psychiatry, part 2: pathogenesis and aetiology. Lancet Psychiatry. 2016 Jan;3(1):84-90. doi: 10.1016/S2215-0366(15)00360-0. Epub 2015 Nov 11. PMID 26573969
- [Background] Stephan KE, Schlagenhauf F, Huys QJM, Raman S, Aponte EA, Brodersen KH, Rigoux L, Moran RJ, Daunizeau J, Dolan RJ, Friston KJ, Heinz A. Computational neuroimaging strategies for single patient predictions. Neuroimage. 2017 Jan 15;145(Pt B):180-199. doi: 10.1016/j.neuroimage.2016.06.038. Epub 2016 Jun 22. PMID 27346545
- [Background] Corlett PR, Fletcher PC. Computational psychiatry: a Rosetta Stone linking the brain to mental illness. Lancet Psychiatry. 2014 Oct;1(5):399-402. doi: 10.1016/S2215-0366(14)70298-6. Epub 2014 Aug 12. No abstract available. PMID 26361002
- [Background] Hasler G. Can the neuroeconomics revolution revolutionize psychiatry? Neurosci Biobehav Rev. 2012 Jan;36(1):64-78. doi: 10.1016/j.neubiorev.2011.04.011. Epub 2011 Apr 29. PMID 21550365
- [Background] Huys QJ, Maia TV, Frank MJ. Computational psychiatry as a bridge from neuroscience to clinical applications. Nat Neurosci. 2016 Mar;19(3):404-13. doi: 10.1038/nn.4238. PMID 26906507
- [Background] Montague PR, Dolan RJ, Friston KJ, Dayan P. Computational psychiatry. Trends Cogn Sci. 2012 Jan;16(1):72-80. doi: 10.1016/j.tics.2011.11.018. Epub 2011 Dec 14. PMID 22177032
- [Background] Keks N, Hope J, Keogh S. Switching and stopping antidepressants. Aust Prescr. 2016 Jun;39(3):76-83. doi: 10.18773/austprescr.2016.039. Epub 2016 Jun 1. PMID 27346915
- [Background] Cipriani A, Furukawa TA, Salanti G, Chaimani A, Atkinson LZ, Ogawa Y, Leucht S, Ruhe HG, Turner EH, Higgins JPT, Egger M, Takeshima N, Hayasaka Y, Imai H, Shinohara K, Tajika A, Ioannidis JPA, Geddes JR. Comparative efficacy and acceptability of 21 antidepressant drugs for the acute treatment of adults with major depressive disorder: a systematic review and network meta-analysis. Lancet. 2018 Apr 7;391(10128):1357-1366. doi: 10.1016/S0140-6736(17)32802-7. Epub 2018 Feb 21. PMID 29477251
- [Background] Koesters M, Ostuzzi G, Guaiana G, Breilmann J, Barbui C. Vortioxetine for depression in adults. Cochrane Database Syst Rev. 2017 Jul 5;7(7):CD011520. doi: 10.1002/14651858.CD011520.pub2. PMID 28677828
- [Background] Hartwig V, Giovannetti G, Vanello N, Lombardi M, Landini L, Simi S. Biological effects and safety in magnetic resonance imaging: a review. Int J Environ Res Public Health. 2009 Jun;6(6):1778-98. doi: 10.3390/ijerph6061778. Epub 2009 Jun 10. PMID 19578460
- [Background] Felice D, Guilloux JP, Pehrson A, Li Y, Mendez-David I, Gardier AM, Sanchez C, David DJ. Vortioxetine Improves Context Discrimination in Mice Through a Neurogenesis Independent Mechanism. Front Pharmacol. 2018 Mar 12;9:204. doi: 10.3389/fphar.2018.00204. eCollection 2018. PMID 29593535
- [Background] Hayakawa YK, Sasaki H, Takao H, Hayashi N, Kunimatsu A, Ohtomo K, Aoki S. Depressive symptoms and neuroanatomical structures in community-dwelling women: A combined voxel-based morphometry and diffusion tensor imaging study with tract-based spatial statistics. Neuroimage Clin. 2014 Mar 12;4:481-7. doi: 10.1016/j.nicl.2014.03.002. eCollection 2014. PMID 24818074
- [Background] Colle R, Dupong I, Colliot O, Deflesselle E, Hardy P, Falissard B, Ducreux D, Chupin M, Corruble E. Smaller hippocampal volumes predict lower antidepressant response/remission rates in depressed patients: A meta-analysis. World J Biol Psychiatry. 2018 Aug;19(5):360-367. doi: 10.1080/15622975.2016.1208840. Epub 2016 Aug 15. PMID 27376473
- [Background] Osimo EF, Pillinger T, Rodriguez IM, Khandaker GM, Pariante CM, Howes OD. Inflammatory markers in depression: A meta-analysis of mean differences and variability in 5,166 patients and 5,083 controls. Brain Behav Immun. 2020 Jul;87:901-909. doi: 10.1016/j.bbi.2020.02.010. Epub 2020 Feb 27. PMID 32113908
- [Background] Kojima M, Matsui K, Mizui T. BDNF pro-peptide: physiological mechanisms and implications for depression. Cell Tissue Res. 2019 Jul;377(1):73-79. doi: 10.1007/s00441-019-03034-6. Epub 2019 May 10. PMID 31076872
- [Background] Ogyu K, Kubo K, Noda Y, Iwata Y, Tsugawa S, Omura Y, Wada M, Tarumi R, Plitman E, Moriguchi S, Miyazaki T, Uchida H, Graff-Guerrero A, Mimura M, Nakajima S. Kynurenine pathway in depression: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2018 Jul;90:16-25. doi: 10.1016/j.neubiorev.2018.03.023. Epub 2018 Mar 30. PMID 29608993
- [Background] Verdonk F, Petit AC, Abdel-Ahad P, Vinckier F, Jouvion G, de Maricourt P, De Medeiros GF, Danckaert A, Van Steenwinckel J, Blatzer M, Maignan A, Langeron O, Sharshar T, Callebert J, Launay JM, Chretien F, Gaillard R. Microglial production of quinolinic acid as a target and a biomarker of the antidepressant effect of ketamine. Brain Behav Immun. 2019 Oct;81:361-373. doi: 10.1016/j.bbi.2019.06.033. Epub 2019 Jun 28. PMID 31255681
- [Background] Harrison NA, Voon V, Cercignani M, Cooper EA, Pessiglione M, Critchley HD. A Neurocomputational Account of How Inflammation Enhances Sensitivity to Punishments Versus Rewards. Biol Psychiatry. 2016 Jul 1;80(1):73-81. doi: 10.1016/j.biopsych.2015.07.018. Epub 2015 Aug 1. PMID 26359113
- [Background] Chen G, Bian H, Jiang D, Cui M, Ji S, Liu M, Lang X, Zhuo C. Pseudo-continuous arterial spin labeling imaging of cerebral blood perfusion asymmetry in drug-naive patients with first-episode major depression. Biomed Rep. 2016 Dec;5(6):675-680. doi: 10.3892/br.2016.796. Epub 2016 Oct 31. PMID 28101340
- [Background] Ota M, Noda T, Sato N, Hattori K, Teraishi T, Hori H, Nagashima A, Shimoji K, Higuchi T, Kunugi H. Characteristic distributions of regional cerebral blood flow changes in major depressive disorder patients: a pseudo-continuous arterial spin labeling (pCASL) study. J Affect Disord. 2014 Aug;165:59-63. doi: 10.1016/j.jad.2014.04.032. Epub 2014 Apr 21. PMID 24882178
- [Background] Cooper CM, Chin Fatt CR, Liu P, Grannemann BD, Carmody T, Almeida JRC, Deckersbach T, Fava M, Kurian BT, Malchow AL, McGrath PJ, McInnis M, Oquendo MA, Parsey RV, Bartlett E, Weissman M, Phillips ML, Lu H, Trivedi MH. Discovery and replication of cerebral blood flow differences in major depressive disorder. Mol Psychiatry. 2020 Jul;25(7):1500-1510. doi: 10.1038/s41380-019-0464-7. Epub 2019 Aug 6. PMID 31388104
- [Background] Kaichi Y, Okada G, Takamura M, Toki S, Akiyama Y, Higaki T, Matsubara Y, Okamoto Y, Yamawaki S, Awai K. Changes in the regional cerebral blood flow detected by arterial spin labeling after 6-week escitalopram treatment for major depressive disorder. J Affect Disord. 2016 Apr;194:135-43. doi: 10.1016/j.jad.2015.12.062. Epub 2016 Jan 21. PMID 26826533
- [Background] Ruckbeil MV, Hilgers RD, Heussen N. Randomization in survival studies: An evaluation method that takes into account selection and chronological bias. PLoS One. 2019 Jun 3;14(6):e0217946. doi: 10.1371/journal.pone.0217946. eCollection 2019. PMID 31158260
- [Background] Montgomery SA, Asberg M. A new depression scale designed to be sensitive to change. Br J Psychiatry. 1979 Apr;134:382-9. doi: 10.1192/bjp.134.4.382. PMID 444788
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Sheehan DV, Harnett-Sheehan K, Spann ME, Thompson HF, Prakash A. Assessing remission in major depressive disorder and generalized anxiety disorder clinical trials with the discan metric of the Sheehan disability scale. Int Clin Psychopharmacol. 2011 Mar;26(2):75-83. doi: 10.1097/YIC.0b013e328341bb5f. PMID 21102344
- [Background] Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995 Jul;167(1):99-103. doi: 10.1192/bjp.167.1.99. PMID 7551619
- [Background] Starkstein SE, Mayberg HS, Preziosi TJ, Andrezejewski P, Leiguarda R, Robinson RG. Reliability, validity, and clinical correlates of apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 1992 Spring;4(2):134-9. doi: 10.1176/jnp.4.2.134. PMID 1627973
- [Background] Brown S, Rittenbach K, Cheung S, McKean G, MacMaster FP, Clement F. Current and Common Definitions of Treatment-Resistant Depression: Findings from a Systematic Review and Qualitative Interviews. Can J Psychiatry. 2019 Jun;64(6):380-387. doi: 10.1177/0706743719828965. Epub 2019 Feb 14. PMID 30763119
- [Background] Friston K, Mattout J, Trujillo-Barreto N, Ashburner J, Penny W. Variational free energy and the Laplace approximation. Neuroimage. 2007 Jan 1;34(1):220-34. doi: 10.1016/j.neuroimage.2006.08.035. Epub 2006 Oct 20. PMID 17055746
- [Background] Daunizeau J, Adam V, Rigoux L. VBA: a probabilistic treatment of nonlinear models for neurobiological and behavioural data. PLoS Comput Biol. 2014 Jan;10(1):e1003441. doi: 10.1371/journal.pcbi.1003441. Epub 2014 Jan 23. PMID 24465198
- [Background] O'Doherty JP, Hampton A, Kim H. Model-based fMRI and its application to reward learning and decision making. Ann N Y Acad Sci. 2007 May;1104:35-53. doi: 10.1196/annals.1390.022. Epub 2007 Apr 7. PMID 17416921
- [Background] Meyniel F, Goodwin GM, Deakin JW, Klinge C, MacFadyen C, Milligan H, Mullings E, Pessiglione M, Gaillard R. A specific role for serotonin in overcoming effort cost. Elife. 2016 Nov 8;5:e17282. doi: 10.7554/eLife.17282. PMID 27824554